CLINICAL TRIAL: NCT04729413
Title: Promoting HIV Health Behaviors Among Pregnant Couples in Zambia Using an Adaptive Relationship Strengthening Intervention
Brief Title: Happy Homes, Healthy Families: A Relationship Strengthening Intervention for Pregnant Couples Affected by HIV in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-1529; R00MH116735-03 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: HIV Infections; Pregnancy Related
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Couples are randomized 1:1 to receive the intervention (couples counseling and health education) or control (enhanced standard of care) in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couples Counseling Intervention (Experimental): Couples in the intervention group will receive two group health education sessions (one during pregnancy and one postpartum) covering information on pregnancy and postpartum health, as well as three couple counseling visits (one during pregnancy and two postpartum). The couples counseling sessions will provide (1) information on key relationship topics (communication, trust and respect, love and support); (2) relationship skills exercises (role playing); and (3) the opportunity to discuss health and relationship priorities/goals of the couple.
  Interventions: Behavioral: Couples Counseling
- Control (Sham Comparator): Couples assigned to the control group will receive two group health education sessions (one during pregnancy and one postpartum) covering information on pregnancy and postpartum health. Couples will also have the opportunity after the trial is complete to opt-in to receive a condensed one-session couples counseling visit (data not to be used for study purposes but offered for ethical reasons).
  Interventions: Other: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Couples Counseling — Psychoeducational counseling on relationships and maternal and child health in the context of HIV.
  Arms: Couples Counseling Intervention
Other: Enhanced Standard of Care — Enhanced standard of care with education on pregnancy and postpartum health, similar to what is presented to women at routine antenatal and postpartum care.
  Other Names: Control/comparator
  Arms: Control

SUMMARY:
The objective of this study is to test the preliminary efficacy of a novel couples' counseling intervention to promote the health of pregnant women living with HIV in Lusaka, Zambia.

DETAILED DESCRIPTION:
The central hypothesis of this study is that women living with HIV in heterosexual couples that have better relationship functioning and more social support will have greater odds of achieving optimal health during and after pregnancy. The study further hypothesizes that the couples-based intervention will improve interpersonal dynamics, such as communication, and in intrapersonal factors, such as women's mental health, which will mediate intervention effects on HIV care and treatment outcomes. The study will test the hypotheses through two specific aims: (1) compare service utilization and prevention of mother-to-child transmission (PMTCT) outcome indicators in two study conditions; and (2) establish the effect of the intervention on intra- and inter-personal mechanisms influencing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual couple in a stable relationship (defined as sleeping under the same roof at least once a week)
* Relationship has lasted ≥ 6 months
* Both partners live in the clinic catchment area and plan to continue residing there for at least six months
* Both partners are at least 18 years of age
* Both partners willing to participate in the intervention
* Female partner is no more than 36 weeks pregnant
* Female partner is diagnosed as HIV-positive
* Severe intimate partner violence (World Health Organization definition) has not occurred within the couple in the past 6 months.

Exclusion Criteria:

* Same-sex couple
* couple who does not sleep under the same roof at least once a week
* Relationship has lasted <6 months
* One or both partners live outside the clinic catchment area
* One or both partners plan to move outside the clinic catchment area
* One or both partners are <18 years of age
* One or both partners unwilling to participate in the intervention
* Female partner is greater than 36 weeks pregnant
* Female partner is HIV-negative
* Severe intimate partner violence (World Health Organization definition) has occurred within the couple in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Female Viral Suppression | Month 6 postpartum
  Laboratory testing of blood samples. A result of <1,000 HIV viral copies/mL indicates viral suppression.

SECONDARY OUTCOMES:
Self-reported 30-day antiretroviral therapy adherence | Month 6 postpartum
  Survey question: "In the last 30 days, on how many days did you miss at least one dose of any of your HIV medicines?" Continuous measurement from 0 days to 30 days.
Self-reported exclusive breastfeeding | Month 6 postpartum
  Survey question: "How is the baby currently being fed?" Exclusive breastfeeding is defined as providing only breastmilk to the infant for the first 6 months of life.
Self-reported postpartum use of family planning | Month 6 postpartum
  Survey question: "Are you currently using any form of family planning?" (yes)
Self-reported infant HIV testing | Month 6 postpartum
  Survey question: "Has the baby been tested for HIV?" (yes)

OTHER OUTCOMES:
Female Viral Suppression | Week 6 postpartum
  Laboratory testing of blood samples. A result of <1,000 HIV viral copies/mL indicates viral suppression.
Self-reported 30-day antiretroviral therapy adherence | Week 6 postpartum
  Survey question: "In the last 30 days, on how many days did you miss at least one dose of any of your HIV medicines?" Continuous measurement from 0 days to 30 days.
Self-reported exclusive breastfeeding | Week 6 postpartum
  Survey question: "How is the baby currently being fed?" Exclusive breastfeeding is defined as providing only breastmilk to the infant for the first 6 months of life.
Self-reported postpartum use of family planning | Week 6 postpartum
  Survey question: "Are you currently using any form of family planning?" (yes)
Self-reported infant HIV testing | Week 6 postpartum
  Survey question: "Has the baby been tested for HIV?" (yes)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hampanda, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Chipata Health Centre, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No